CLINICAL TRIAL: NCT00787540
Title: Chest Pain, Illness Perception Compliance and Psychosocial Outcome After Coronary Arteriography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Ali Shalabi, Hillel Yaffe Medical Center
Other Study IDs: 0051-08 HYMC
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Coronary Disease
Keywords: Coronary disease; Psychosocial; Nursing
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- I: Coronary Slow Flow Patients
- II: Coronary Artery Occlusion Patients

SUMMARY:
Chest pain, illness perception compliance and psychosocial outcome after coronary arteriography. A comparison between patients which were diagnosed with slow coronary flow and patients who have been diagnosed with coronary artery occlusion. We hope to prove that the more knowledge and awareness the patient has about his disease the better his compliance and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with slow flow or coronary artery occlusion

Exclusion Criteria:

* All other patients

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the coronary unit at the Hillel Yaffe Medical Center, Hadera, Israel
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Coronary Care Unit, Heart Institute, Hillel Yaffe Medical Center, Hadera, Israel